CLINICAL TRIAL: NCT02754388
Title: Early Detection of Lung Cancer With Low-dose Multislice Computed Tomography (LDCT)- a Screening Program
Brief Title: Early Detection of Lung Cancer With Low-dose Multislice Computed Tomography
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201512060RIND
Record Dates: First submitted 2016-04-10; First posted 2016-04-28 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
Keywords: LDCT, screening, health behavior, psychological factors
MeSH Terms: conditions — Lung Neoplasms; Health Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
Lung cancer is one of the leading causes of cancer-related death in Taiwan. Early diagnosis of lung cancer may improve cancer survival. Low-dose computed tomography (LDCT) was thought to be the best screening tool for lung cancer. However, there is growing concerns about radiation exposure, high cost, and high rate of false-positive screening result. Epidemiologic studies from western countries showed that cigarette smoking is the major cause of lung cancer, and other risk factors may include age, environmental pollution, occupational exposures (included of radon exposure), gender, race, and pre-existing lung diseases. Adenocarcinoma is the major type of lung cancer in Taiwan and is less attributable to smoking. The investigators need a different risk prediction model adapted to the investigators country.

National Taiwan University Hospital Chu-Tung Branch initiated the lung cancer screening by LDCT since June 2015. Many people can get the LDCT screening with affordable price with the subsidy from enterprise donation. The purpose of this study is observing those participants with 2-year follow-up. Furthermore, those data may connect with another study of "Low dose computed tomography screening study in nonsmoker with risk factors for lung cancer in Taiwan" （Non-smoker study）which is implemented in other hospitals in Taiwan.For reality limiting, After one year, the enrollment rate was a lot lower than expected. We extended the enrollment time but only observe those participants for one year not two year..

DETAILED DESCRIPTION:
Lung cancer is one of the leading causes of cancer-related death in Taiwan. Early diagnosis of lung cancer may improve cancer survival. Low-dose computed tomography (LDCT) was thought to be the best screening tool for lung cancer. However, there is growing concerns about radiation exposure, high cost, and high rate of false-positive screening result. Epidemiologic studies from western countries showed that cigarette smoking is the major cause of lung cancer, and other risk factors may include age, environmental pollution, occupational exposures (included of radon exposure), gender, race, and pre-existing lung diseases. Adenocarcinoma is the major type of lung cancer in Taiwan and is less attributable to smoking. The investigators need a different risk prediction model adapted to the investigators country.

National Taiwan University Hospital Chu-Tung Branch initiated the lung cancer screening by LDCT since June 2015. Many people can get the LDCT screening with affordable price with the subsidy from enterprise donation. The purpose of this study is observing those participants with 2-year follow-up. Furthermore, those data may connect with another study of "Low dose computed tomography screening study in nonsmoker with risk factors for lung cancer in Taiwan" （Non-smoker study）which is implemented in other hospitals in Taiwan.

Aim 1: Being the control group of the non-smoker study, the investigators collect the relevant information from participants to validate and modify their risk assessment model. Applying the same the questionnaires of the non-smoker study and results of LDCT screening in different population. All data could provide extra information to improve their risk prediction model for predicting lung cancer in non-smokers in Taiwan.

Aim 2: To establish the local epidemiological data for lung pathology. From the baseline data, screening results of LDCT, telephone follow up on questionable lesions, collection of patient's medical records, and linkage to National Health Insurance Database, the investigators will be able to establish local epidemiology data on lung pathology as well as information on screening accuracy of LDCT.

Aim 3: To examine the psychosocial impacts and health behaviors of the participants receiving LDCT. Questionnaire surveys provide the understanding of anxiety and life quality at several time points since LDCT screening. The study was to investigate whether the screening results were associated with health behaviors change, such as smoking, drinking, and exercise.

With low enrollment rate in first year, we decided to extend the enrollment period. But we only observed those participants for one year, not 2 year. So far we carry on the analysis and the discussion.

Keywords: Lung cancer, Low dose computed tomography, screening, health behavior, psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* age>=20
* self pay the LDCT in National Taiwan University Hospital Chu-Tung Branch
* ability to understand the informed consent form for complete the questionnaires
* be willing and able to accept telephone access at the time scheduled

Exclusion Criteria:

NA

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients received LDCT screening at NTUH Chu-Tung Branch
Sampling Method: Non-Probability Sample
Enrollment: 1334 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Abnormal ct finding detection rate | 1-month
  Abnormal ct finding detection rate is defined as number of abnormal ct finding/total enroll number

SECONDARY OUTCOMES:
Change in Chinese 14-item Perceived Stress Scale (Chinese 14-item PSS) score | 6-month
  Stress will be measured using the Chinese 14-item Perceived Stress Scale (Chinese 14-item PSS) at baseline and 6 month follow-up.
Change in Chinese Health Questionnaire-12 (CHQ-12) score | 12-month
  Psychological morbidity will be measured using the Chinese Health Questionnaire (CHQ-12) at baseline and 12 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, MD, PhD, Principal Investigator — National Taiwan University Hospital Chu-Tung Branch

IPD SHARING:
Plan to Share IPD: No